CLINICAL TRIAL: NCT06125925
Title: Catheter Ablation in Atrial Fibrillation Patients With Heart Failure With Preserved Ejection Fraction: an International, Prospective, Multi-center, Randomized Controlled Study (STABLE-SR IV Trial)
Brief Title: Catheter Ablation in Atrial Fibrillation Patients With HFpEF (STABLE-SR IV Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Minglong Chen, Director of Heart Center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-SR-659
Record Dates: First submitted 2023-10-13; First posted 2023-11-09 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: atrial fibrillation; HFpEF; radiofrequency catheter ablation; drug therapy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The End Point and Adverse Event Committee is constituted of three experts in the field of heart failure and ablation of atrial fibrillation, but independent of the study. The End Point Adverse Event Committee have received blinded data regarding all serious adverse events, all deaths, all hospitalizations, all outpatient or emergency visits, all cerebrovascular accidents, and all first recurrences of atrial fibrillation, from the Contact Research Organization. The End Point and Adverse Event Committee was responsible for the classification of all received events, for the determination of which events fulfill the end point criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency catheter ablation (RFCA) (Experimental): Radiofrequency ablation is adopted in the study, instead of cryo ablation, surgical ablation or pulsed field ablation. 3-dimensional model is constructed after transseptal puncture. Circumferential pulmonary vein isolation (CPVI) is performed with irrigated contact force catheter. Previously published STABLE-SR approach is recommended as the ablation strategy beyond CPVI.
  Interventions: Procedure: Radiofrequency catheter ablation (RFCA)
- Medical therapy (Active Comparator): AADs should be prescribed according to the current guidelines, such as amiodarone, dronedarone, or propafenone. In brief, rhythm control is preferred, including electric cardioversion. However, rate control should be considered if rhythm control is contraindicated, intolerated or unpreferred by patients.
  Interventions: Drug: Medical Therapy

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation (RFCA) — Radiofrequency ablation is adopted in the study, instead of cryo ablation, surgical ablation or pulsed field ablation. 3-dimensional model is constructed after transseptal puncture. Circumferential pulmonary vein isolation (CPVI) is performed with irrigated contact force catheter. Previously published STABLE-SR approach is recommended as the ablation strategy beyond CPVI.
  Arms: Radiofrequency catheter ablation (RFCA)
Drug: Medical Therapy — AADs should be prescribed according to the current guidelines, such as amiodarone, dronedarone, or propafenone. In brief, rhythm control is preferred, including electric cardioversion. However, rate control should be considered if rhythm control is contraindicated, intolerated or unpreferred by patients.
  Arms: Medical therapy

SUMMARY:
To investigate whether RFCA is superior to AADs in AF patients with HFpEF on the basis of optimized anti-heart-failure drug therapy regarding their longterm clinical outcomes.

DETAILED DESCRIPTION:
Background: Atrial Fibrillation (AF) is a common cardiac rhythm disorder and radiofrequency catheter ablation (RFCA) has become the first-line therapy in the symptomatic AF patients. Heart failure is often the sister disease with AF. Recently, RFCA was found to be superior to antiarrhythmic drugs (AADs) in heart failure patients with AF and reduced ejection fraction (HFrEF), regarding all-cause mortality and hospitalization for worsening heart failure (HF). However, in heart failure patients with AF and preserved ejection fraction (HFpEF), it remains unknown whether RFCA is superior to AADs in an even larger population, despite several nonrandomized retrospective studies. Thus, this prospective, multi-center, randomized controlled trial aims to investigate whether RFCA could better improve the clinical outcome of AF patients with HFpEF than longterm AADs use.

Aim of this study: To investigate whether RFCA is superior to AADs in AF patients with HFpEF on the basis of optimized anti-heart-failure drug therapy regarding their longterm clinical outcomes.

Design: The STABLE-SR-IV trial is an international, prospective, multi-center, randomized controlled trial. In this trial, physical examination, echocardiogram, NT-proBNP and other blood test would be assessed before enrollment. Those who conform to all the inclusion criteria and absent from any exclusion criteria would enter into a run-in period of 5 weeks (±7 days). Anticoagulation and anti-heart-failure therapy for HFpEF must be optimized according to the current guideline. After the run-in period, inclusion and exclusion criteria would be reassessed. Thereafter, all the subjects enrolled would be randomized into RFCA arm and Medical Therapy arm with a 1:1 manner, namely 218 subjects in each arm. Each arm will follow the protocol of RFCA and medical therapy, respectively. Follow-up duration of this study is up to 2~3 years (12 month enrollment).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal or persistent atrial fibrillation
* CHADS2-VASc score≥ 2
* Conform to the diagnosis of HFpEF

  1. NYHA II-IV level;
  2. Left ventricular ejection fraction (LVEF)≥ 50%;
  3. NT-proBNP≥ 300 pg/mL under sinus rhythm or NT-proBNP≥ 600 pg/mL under atrial fibrillation or flutter;
  4. Evidence of left ventricular diastolic dysfunction/raised left ventricular filling pressure on echocardiogram.
* Sign informed consent

Exclusion Criteria:

* A life expectancy below 2 years due to any non-cardiovascular condition
* Reversible atrial fibrillation, such as hyperthyroidism or hypokalemia-related atrial fibrillation
* Prior atrial fibrillation ablation
* Left atrial size≥ 55 mm
* Heart failure due to any of the following: known genetic hypertrophic cardiomyopathy, infiltrative cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, constrictive pericarditis, active myocarditis, cardiac tamponade, or uncorrected primary valvular disease
* Previous cardiac transplantation, complex congenital heart disease, rheumatic heart disease
* Any contraindication for radiofrequency catheter ablation, antiarrhythmic drugs or anticoagulation
* Acute coronary syndrome, cardiac surgery, angioplasty or cerebrovascular accident within 12 weeks before enrollment
* Severe hepatic and renal dysfunction
* Body mass index> 50 kg/m2
* Female in period of pregnancy or breast-feeding
* Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study
* Involved in other studies

The inclusion and exclusion criteria would be reassessed after run-in period and the cut-off of NT-proBNP would be set as >125 pg/ml under sinus rhythm or >365 pg/ml under AF/atrial flutter (AFL).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of worsening heart failure requiring unplanned hospitalizations or urgent visits, and cardiovascular death (Time-to-first event analysis) | From randomization until completion of the planned follow-up, up to 36 months

SECONDARY OUTCOMES:
Time to hospitalization or urgent visits for heart failure | From randomization until completion of the planned follow-up, up to 36 months
  Worsening heart failure includes worsening heart failure requiring unplanned hospitalization and worsening heart failure requiring urgent visits.
Time to hospitalization for heart failure | From randomization until completion of the planned follow-up, up to 36 months
  In addition to signs and symptoms of HF, the patient should also receive treatment specifically directed at HF, including at least 1 of the following: 1) significant augmentation in oral diuretic therapy; 2) initiation of intravenous diuretic (even a single dose) or vasoactive agent (eg, vasodilator, vasopressor, or inotropic therapy); or 3) mechanical circulatory support or fluid removal.
  Unplanned hospitalization is defined as any unscheduled hospital admission with a length of stay that either exceeds 24 h or crosses a calendar day, and not planned by the investigators. In case the hospitalization is classified as planned by the Investigator and the time interval between the decision to admit and the admission is less than 24 hours, the End Point and Adverse Event Committee will give final classification concerning planned or unplanned.
Time to urgent visits for heart failure | From randomization until completion of the planned follow-up, up to 36 months
  Worsening of Heart Failure Requiring Unplanned Urgent Visits Patients have an urgent, unscheduled office or emergency visit for HF with signs, symptoms, and diagnostic testing results identical to those already described for an HF hospitalization. The patient must also (with the exception of significant augmentation in oral diuretic therapy) require therapy similar to that previously described for an HF hospitalization.
Time to cardiovascular death | From randomization until completion of the planned follow-up, up to 36 months
  All deaths due to cardiovascular reasons and all heart transplants because of terminal HF. Deaths due to worsening of HF, acute coronary syndrome, cerebrovascular accident.
Time to all-cause death | From randomization until completion of the planned follow-up, up to 36 months
  All deaths were reviewed and adjudicated by the Clinical Events Committee
Time to cardiovascular hospitalization | From randomization until completion of the planned follow-up, up to 36 months
  Unplanned Hospitalization due to Cardiovascular Reasons Any in-hospital stay over one date change due to cardiovascular reason, which includes worsening of HF, acute coronary syndrome, cerebrovascular accidents, or other cardiovascular events, and not planned by the investigator. In case the hospitalization is classified as planned by the investigator, and the time interval between the decision to hospitalize and the hospitalization is less than 24 hours, the End Point and Adverse Event Committee will give final classification concerning planned or unplanned.
Total number of worsening heart failure events and cardiovascular deaths | From randomization until completion of the planned follow-up, up to 36 months
Change in quality of life - KCCQ score | Baseline, 3 months, 12 months
  KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ Total Symptom Score incorporates the symptom domains into a single score. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in quality of life - MLWHFQ | Baseline, 3 months, 12 months
  The Mayo AF-Specific Symptom Inventory (MAFSI) is a questionnaire comprised of a 10-item AF symptom checklist that asked about both the frequency and severity of each symptom. MAFSI frequency of symptoms over the past month was recorded as 0 (never), 1 (rarely), 2 (sometimes), 3 (often), and 4 (always) for each of the 10 items listed in the questionnaire. The 10 item responses were summed for a total Frequency Score that ranged from 0 (no AF symptoms) to 40 (worst score).
Change in 6-minute walk test from baseline to Month 3 and Month 12 | Baseline, 3months, 12 months
  The 6-minute walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance.
Change in H2FPEF score from baseline to Month 3 and Month 12 | Baseline, 3 months, 12 months
  The H2FPEF score is a clinical scoring system used to assess the likelihood of heart failure with preserved ejection fraction (HFpEF) in patients with suspected heart failure. It helps in differentiating HFpEF from other causes of dyspnea. The total score ranges from 0 to 5, with higher scores indicating a greater likelihood of HFpEF.
Change in N-terminal pro-B type natriuretic peptide (NT-proBNP) from baseline to Month 3 and Month 12 | Baseline, 3 months, 12 months
  Elevated levels of NT-pro BNP are indicative of increased cardiac stress and can help in the diagnosis, assessment, and monitoring of heart failure.
Change in NYHA class from baseline to Month 3, 6 and 12 | Baseline, 3 months, 12 months
  NYHA class is a widely used system for assessing the functional status and severity of heart failure symptoms in patients, with NYHA class IV being the worst.
Time to change of diuretics | From randomization until completion of the planned follow-up, up to 36 months
  Based on status of baseline diuretics, the intention to treat population will be divided into patients with baseline diuretics and patients without.
  For patients without the usage of baseline diuretics, the outcome of changes in diuretics is the initiation of diuretics during the follow-up period.
  For patients without the usage of baseline diuretics, the outcomes including:
  1. permanent discontinuation;
  2. escalation defined as increased dosage, iv fused diuretic or combination with another diuretic;
  3. de-escalation (including permanent discontinuation or decrease in dosage); Changes in diuretic therapy are analyzed in a time-to-first event fashion using a multivariable Cox regression model to obtain hazard ratios (HRs) and 95% confidence intervals (CIs).
Change in atrial fibrillation burden | Baseline, 12 months
  Atrial fibrillation burden refers to the amount of time that a person with atrial fibrillation spends in an irregular heart rhythm over a specific period, using a Holter monitor.
Time to Atrial Fibrillation recurrence (RFCA arm) | From randomization until completion of the planned follow-up, up to 36 months
  A 30-second episode of AF in ablation group following the 90 day blanking period, confirmed through blinded review by an ECG Core Lab Committee was used for defining the endpoint of recurrent AF.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No